CLINICAL TRIAL: NCT05264883
Title: Comparing the Efficacy and Safety of Venetoclax Combined With Decitabine/Azacitidine and Aclarubicin Versus Venetoclax Combined With Decitabine/Azacitidine in Treatment-Naive Elderly Patients With Acute Myeloid Leukemia
Brief Title: Venetoclax+HMA+Aclarubicin Versus Venetoclax+HMA in Treatment-Naive Elderly Patients With AML
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: The Affiliated Jiangning Hospital of Nanjing Medical University (Other); Huai'an First People's Hospital (Other); Yancheng First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-SR-278
Record Dates: First submitted 2022-02-27; First posted 2022-03-03 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Venetoclax combined with Decitabine/Azacitidine and Aclarubicin (Experimental): Venetoclax (Ven): oral once daily (100 mg d1, 200 mg d2, 400 mg d3-28);
  Decitabine (DAC): 20mg/m2 intravenous for 1 hour daily (d1 to d5);
  Azacitidine (AZA): 75mg/m2 subcutaneous at two different sites daily (d1 to d7);(Choose decitabine or azacitidine according to the patient's wishes)
  Aclarubicin (Acla): 10mg/m2 intravenous daily (d1 to d3);
  Interventions: Drug: Venetoclax-Decitabine/Azacitidine-Aclarubicin Association
- Venetoclax combined with Decitabine/Azacitidine (Active Comparator): Venetoclax (Ven): oral once daily (100 mg d1, 200 mg d2, 400 mg d3-28);
  Decitabine (DAC): 20mg/m2 intravenous for 1 hour daily (d1 to d5);
  Azacitidine (AZA): 75mg/m2 subcutaneous at two different sites daily (d1 to d7);(Choose decitabine or azacitidine according to the patient's wishes)
  Interventions: Drug: Venetoclax-Decitabine/Azacitidine Association

INTERVENTIONS:
Drug: Venetoclax-Decitabine/Azacitidine-Aclarubicin Association — Treatment with Venetoclax+Decitabine/Azacitidine+Aclarubicin
  Arms: Venetoclax combined with Decitabine/Azacitidine and Aclarubicin
Drug: Venetoclax-Decitabine/Azacitidine Association — Treatment with Venetoclax+Decitabine/Azacitidine
  Arms: Venetoclax combined with Decitabine/Azacitidine

SUMMARY:
This research is being done to assess the therapeutic efficacy and safety of a promising regimen (Venetoclax combined with Decitabine/Azacitidine and Aclarubicin) versus Venetoclax combined with Decitabine/Azacitidine in treatment-naive elderly patients with Acute Myeloid Leukemia.

This study involves the following:

Venetoclax, Decitabine/Azacitidine, Aclarubicin (investigational combination) Venetoclax and Decitabine/Azacitidine (per standard of care)

DETAILED DESCRIPTION:
This is an open-label, multicenter, phase Ⅲ randomized clinical trial to compare the therapeutic efficacy and safety of Venetoclax combined with Decitabine/Azacitidine and Aclarubicin versus Venetoclax combined with Decitabine/Azacitidine in treatment-naive elderly patients with Acute Myeloid Leukemia (AML).

The FDA has approved the combination therapy of Venetoclax and Decitabine/Azacitidine for elderly (> 60-year-old) patients with newly diagnosed AML not eligible for intensive chemotherapy. Venetoclax is an inhibitor of BCL-2 (B-cell lymphoma 2, a protein that initiates tumor growth, disease progression, and drug resistance), which can lead to cancer cell death.

Aclarubicin (Acla) is an anthracycline antitumor drug and is a type II topoisomerase Inhibitor that prevents topoisomerase II from binding to DNA primarily by intercalating into DNA strands, resulting in chromatin damage injury without causing DNA damage. In addition to causing chromatin damage, Acla also results in epigenetic inheritance Changes in gene transmission, DNA damage response signals, and apoptosis. Furthermore, in the cytoplasm, Acla can also exert cytotoxic effects by affecting mitochondrial respiratory function. Therefore, Acla is a highly efficient and broad-spectrum chemotherapeutic drug, which is widely used in the treatment of various hematological tumors and solid tumors. In treatment-naive elderly patients with AML, the DCAG (Decitabine-Cytarabine-Aclarubicin-GCSF) regimen can improve the prognosis according to our previous research results. Acla also has relatively mild side effects in the treatment of AML patients.

Participants will be randomly assigned to one of the different treatment groups and followed with consolidated therapy with the same regimen of 2-4 cycles. After completion of study treatment, participants are followed up every 3 months for up to 2 years.

It is expected that about 170 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute myeloid leukemia (AML) diagnosed by bone marrow morphology and immunophenotyping (in line with WHO 2016 diagnostic criteria);
2. No previous anti-acute leukemia treatment (including demethylating drugs), except hydroxyurea and Leukocyte apheresis;
3. Exclude acute promyelocytic leukemia (APL) at the bone marrow morphology or molecular level;
4. Age 60-80 years old;
5. Aspartate aminotransferase (ALT), alanine aminotransferase (AST), and alkaline phosphatase (ALP)≤ 3×upper limit of normal (ULN), serum bilirubin≤ 1.5×ULN; serum creatinine≤ 2.0×ULN; serum heart rate≤ 2.0×ULN;
6. LVEF determined by echocardiography≥ 50%;
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2;
8. Obtain informed consent signed by the patient or legal representative.

Exclusion Criteria:

1. Acute promyelocytic leukemia, myeloid sarcoma, accelerated phase and blast of chronic myeloid leukemia;
2. Patients with relapsed AML;
3. Allergy to any drug involved in the program;
4. Pregnant, lactating women and patients of childbearing age who are unwilling to take contraceptive measures;
5. The liver and kidney functions are obviously abnormal, exceeding the inclusion criteria;
6. Structural heart disease, such as uncontrolled or symptomatic arrhythmia, congestive heart disease, heart failure or myocardial infarction within 6 months prior to screening, resulting in clinical symptoms or abnormal cardiac function;
7. Suffering from other malignant tumors at the same time; except for the following cases: ①Have received treatment for the purpose of cure, and have no known active malignance for ≥5 years before enrollment; ② Adequately treated non-melanoma skin cancer or malignant lentigo with no signs of disease (even if less than 3 years before randomization); ③ Adequately treated carcinoma in situ with no signs of disease (even if less than 3 years before randomization);
8. AIDS patients, syphilis patients, active type Hepatitis B (HBV-DNA detectable) patients, and Hepatitis C patients;
9. Any concurrent medical condition or disease (such as active systemic infection) that may interfere with study procedures or results, or which, in the judgment of the investigator, poses a risk to participation in this study；
10. Inability to understand or comply with the research protocol;
11. Received major surgery within 4 weeks before randomization;
12. Participate in other clinical investigators at the same time one month before enrollment.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-06-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with complete remission (CR) and complete remission with incomplete marrow recovery (CRi) | From randomization to the end of Cycle 1 (each cycle is 28 days)
  CR is defined as absolute neutrophil count > 10^9/ L, platelets > 100×10^9/L, red cell transfusion independence, and bone marrow with < 5% blasts. CRi is defined as bone marrow with less than 5% blasts, and absolute neutrophils of < 10^9/L or platelets < 100×10^9/L.

SECONDARY OUTCOMES:
Partial Remission (PR) Rate | From randomization to the end of Cycle 1 (each cycle is 28 days)
  PR is defined as bone marrow with 5%~25% blasts, at least 50% lower than the initial diagnosis.
Overall Response Rate (ORR) | From randomization to the end of Cycle 1 (each cycle is 28 days)
  Complete Remission/ Complete Remission with incomplete count recovery/ Partial Remission/ Morphologic Leukemia Free State
Rate of Minimal Residual Disease (MRD) negativity | From randomization to the end of Cycle 1 (each cycle is 28 days)
  Percentage of participants who converted to MRD < 10^-3 before initiation of consolidation therapy. MRD is measured by MFC and RT-qPCR.
Overall survival (OS) | From the time of randomization to time for up to 2 years
  It is measured from the date of randomization to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.
Disease-Free Survival (DFS) | From the time of randomization to time for up to 2 years
  It is defined as the time from the date of CR/CRi to the date of recurrence or death.
Early Mortality Rate | From the time of randomization to time for up to 2 years
Cumulative incidence of relapse (CIR) | From the time of CR/CRi to time for up to 2 years
  It is measured from the date of CR/CRi to the date of relapse.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No